CLINICAL TRIAL: NCT00244439
Title: A Multi-Center Phase III Study to Evaluate MALG, a Novel Malathion 0.05%Formulation, for the Control of Head Lice in Pediatric and Adult Subjects With Pediculosis Capitis
Brief Title: Safety and Efficacy of a Novel Malathion Formulation in the Treatment of Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Medical Director, Taro Pharmaceuticals USA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MALG-0506
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Lice Infestations
Keywords: Head Lice; Pediculosis capitis
MeSH Terms: conditions — Lice Infestations | interventions — Malathion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MALG
  Interventions: Drug: MALG
- 2 (Active Comparator): Ovide
  Interventions: Drug: Ovide (malathion) lotion 0.05%
- 3 (Active Comparator): Permethrin 1%
  Interventions: Drug: Permethrin 1%

INTERVENTIONS:
Drug: MALG — 30 minute application
  Arms: 1
Drug: Ovide (malathion) lotion 0.05% — 8-12 hour application
  Arms: 2
Drug: Permethrin 1% — 10 minute application
  Arms: 3

SUMMARY:
Current treatments for head lice include over-the-counter products such as permethrin and prescription products such as OVIDE (malathion 0.5%) lotion. In a previous phase II study, a novel, easy-to-use malathion 0.5% formulation was found to be a safe treatment for head lice. The current study will compare the efficacy and safety of this novel formulation of malathion with OVIDE and with an over-the-counter permethrin product.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active head lice infestation
* Patient, parent or guardian must be able to apply the treatment
* Entire household must be screened
* All infested persons must agree to participate

Exclusion Criteria:

* Allergy to pediculicides, hair care products or chrysanthemums
* Scalp conditions other than head lice
* Previous head lice treatment within the past 4 weeks
* Female patients who are pregnant or nursing

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2005-12; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Cure of Head Lice | 4 weeks

SECONDARY OUTCOMES:
Safety of treatments | 4 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Investigator Site, Scottsdale, Arizona
  - Investigator Site, Miami, Florida
  - Investigator Site, St. Petersburg, Florida
  - Investigator Site, West Palm Beach, Florida
  - Investigator Site, New York, New York
  - Investigator Site, Miamiville, Ohio